CLINICAL TRIAL: NCT05394454
Title: The Effect of Non-invasive Bladder Stimulation Technique on Collecting Urine Specimen in Infants Under One Year Old: Randomized Controlled Trial
Brief Title: The Effect of Non-invasive Bladder Stimulation Technique on Collecting Urine Specimen in Infants Under One Year Old
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nihan Korkmaz, Research assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Barış090221
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Urine Specimen Collection
Keywords: urine specimen; infant; bladder stimulation; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): * Breast milk/formula milk/water intake appropriate for the infant's age and weight will be provided 20-30 minutes before collecting the urine sample.
  * Before the procedure, the infant's heart rate, saturation and Flacc scale score (by the researcher and the observer nurse) will be recorded.
  * Genital area will be cleaned.
  * Infants will be held under the armpit by a parent, baby boys will be held with their legs hanging down, and baby girls will be held in hip flexion position.
  * Infants with spontaneous voiding during the period from the beginning of the research procedure until the infant is positioned will be excluded from the study.
  * The bladder stimulation technique will be repeated sequentially for 3 minutes until micturition begins.
  * After the maneuvers are started, the infants's heart rate and saturation FLACC pain scale score will be recorded at the 1st and 3rd minutes.
  * The success of the procedure and the duration of the procedure will be recorded
  Interventions: Procedure: Bladder stimulation technique
- Control Group (No Intervention): * Breast milk/formula milk/water intake appropriate for the infant's age and weight will be provided 20-30 minutes before collecting the urine sample.
  * Before the procedure, the infant's heart rate, saturation and Flacc scale score (by the researcher and the observer nurse) will be recorded.
  * Genital area will be cleaned.
  * Infants will be held under the armpit by a parent, baby boys will be held with their legs hanging down, and baby girls will be held in hip flexion position.
  * Infants with spontaneous voiding during the period from the beginning of the research procedure until the infant is positioned will be excluded from the study.
  * Bladder stimulation technique will not be applied.
  * Infants will be observed for 3 minutes. Infants's heart rate and saturation FLACC pain scale score will be recorded at the 1st and 3rd minutes.
  * The success of the procedure and the duration of the procedure will be recorded

INTERVENTIONS:
Procedure: Bladder stimulation technique — The bladder stimulation technique consists of two consecutive maneuvers. In the first maneuver, the bladder is stimulated by tapping the suprapubic region for 30 seconds at a frequency of 100 touches per minute. In the second maneuver, circular massage is applied to the paravertebral region for 30 seconds. The two stimulation maneuvers will be repeated alternately for 3 minutes (180 seconds) until micturition begins.
  Arms: Experimental Group

SUMMARY:
Urinary tract infection (UTI) is common in early childhood. The American Academy of Pediatrics accepts suprapubic aspiration and bladder catheterization as the gold standard for the diagnosis of UTI. However, these techniques are painful and invasive. Clean-caught urine provides an acceptable urine specimen for the diagnosis of UTI, although this method is possible for toilet-trained children. Bladder stimulation maneuvers that allow clean-caught urine specimens have recently been identified in children who are not toilet trained. This study was planned to examine the effect of non-invasive bladder stimulation technique used in collecting urine specimen in infants under the age of one, on the success of the procedure, the duration of the procedure, the physiological parameters of the baby, and the level of pain.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is a common bacterial infection in early childhood (Morello et al 2016). UTI symptoms in infants are nonspecific. Therefore, it is important to take a good urine specimen for diagnosis. In practice, different techniques are used to collect urine specimen. These techniques are suprapubic aspiration, urinary catheterization, sterile urine collection bag, and cleanly caught urine. The American Academy of Pediatrics (AAP) recommends collecting urine specimen by suprapubic aspiration (SPA) and urinary catheterization methods for the diagnosis of UTI. The sterile urine collection bag is a non-invasive urine collection technique. This technique is both time consuming and the urine obtained has high bacterial contamination. (Kaufman 2020). Clean-caught urine provides an acceptable urine specimen for the diagnosis of UTI. However, this technique is possible for toilet-trained children (Roberts et al. 2016).

Recently, Herreros Fernández et al. (2013) described a clean-caught urine collection technique based on bladder stimulation and lumbar paravertebral massage. This technique was successful in 86% of newborns, with an average duration of 57 seconds.

When the literature is reviewed, more evidence is needed regarding the bladder stimulation technique in children without toilet training. Examining the effects of parasympathetic system stimulating maneuvers on children's physiological parameters and pain will contribute to more knowledge about the technique.

This study will be conducted to investigate the effect of non-invasive bladder stimulation technique on the success of the procedure, the duration of the procedure, the physiological parameters and the level of pain in collecting urine specimens in infants under the age of one.

Study Population and Sampling: The study population will consist of infants without toilet training, who applied to the Pediatric Emergency Service of a university hospital and whose urine specimen should be collected for diagnostic purposes.The sample of the study will consist of 64 infants (Experimental group=32, Control group=32) under the age of one who applied to the Pediatric Emergency Service of a university hospital, met the criteria for inclusion in the study, and received written consent from their parents. In calculating the sample size, Altuntaş et al. (2015) benefited from the study. Considering the success rates; The minimum number of samples to be taken was determined as 64 (Experimental group=32, Control group=32) with 95% confidence (1-α), 95% test power (1-β), w=0.453 effect size.

Randomization: Infants who meet the research sample selection criteria will be assigned to the experimental and control groups using the balanced block randomization method. Tran et al (2016) reported increasing age in children as a factor affecting the success of the procedure. For this reason, the block randomization method will be preferred in order to ensure that the infants are distributed homogeneously according to the age groups. In order to assign infants to the experimental and control groups, 4 blocks will be created on the computer (www.random.org) according to age (1-3 months, 4-6 months, 7-9 months, 10-12 months). Each block will contain 16 (8 experimental, 8 control) babies.

Data Collection Method The data will be collected by the researcher in the unit where the study is planned to be carried out.

Data Collection Tools

Data Collection Form: Prepared by the researcher. The form includes questions about the infant's age, weight, gender, whether he is circumcised if male, fever, heartbeat, saturation level, FLACC scale score, and procedure success and duration of the procedure.

The FLACC Pain Scale was developed by Merkel et al in 1997. Five behavioral parameters are evaluated on the FLACC scale. Each of the baby's facial expression, leg movements, activity, crying, and comfortability parameters take the value 0, 1, 2. The total score is between 0 and 10 (Merkel et al. 1997). The Turkish validity and reliability of the scale was performed by Şenaylı et al.(2006).

Pulse Oximeter Device to detect the oxygen saturation (SPO2) and heart rate (HR) of infants before, during and after the procedure

Intervention

The bladder stimulation technique consists of two consecutive maneuvers. In the first maneuver, the bladder is stimulated by tapping the suprapubic region for 30 seconds at a frequency of 100 touches per minute. In the second maneuver, circular massage is applied to the paravertebral region for 30 seconds. The two stimulation maneuvers will be repeated alternately for 3 minutes (180 seconds) until micturition begins. Maneuvers will be performed by the researcher. Infants in both groups will be held under the armpit by a parent, male infants will be held in the drooping legs, and female infants will be held in the hip flexion position. Bladder stimulation technique will be applied to the experimental group, but not to the control group.

Interventions to be applied to the experimental group:

* Breastmilk/formula milk/water intake appropriate for the infant's age and weight will be provided 20-30 minutes before the urine specimen is taken.
* Before the procedure, information about the infant in the data collection form will be recorded.
* Before the procedure, the infant 's heart rate, saturation level and Flacc scale score will be recorded. Scoring of the FLACC pain scale will be done by the researcher and a nurse who is not part of the research team.
* Genital area will be cleaned before taking urine specimen.
* İnfant will be held under the armpit by a parent, baby boys will be held with their legs hanging down, and baby girls will be held in hip flexion position.
* Infants with spontaneous voiding during the period from the beginning of the research procedure until the infant is positioned will be excluded from the study. Instead of the infant excluded, the first infant who met the inclusion criteria of the study and presented to the emergency department will be included.
* The bladder stimulation technique consists of two consecutive maneuvers. In the first maneuver, the bladder is stimulated by tapping the suprapubic region for 30 seconds at a frequency of 100 touches per minute. In the second maneuver, circular massage is applied to the paravertebral region for 30 seconds. The two stimulation maneuvers will be repeated alternately for 3 minutes (180 seconds) until micturition begins.
* After the maneuvers are started, the infant will be evaluated with the FLACC pain scale at the 1st and 3rd minutes by the researcher and a nurse who is not part of the research team.
* Heart rate and saturation will be recorded at the 1st and 3rd minutes after the maneuvers are started.
* The success of the procedure and the duration of the procedure will be recorded

Interventions to be applied to the control group:

* Breastmilk/formula milk/water intake appropriate for the infant 's age and weight will be provided 20-30 minutes before the urine specimen is taken.
* Before the procedure, information about the infant in the data collection form will be recorded.
* Before the procedure, the infant's heart rate, saturation level and Flacc scale score will be recorded. Scoring of the FLACC pain scale will be done by the researcher and a nurse who is not part of the research team.
* Genital area will be cleaned before taking urine specimen.
* Infant will be held under the armpit by a parent, baby boys will be held with their legs hanging down, and baby girls will be held in hip flexion position.
* Infant with spontaneous voiding during the period from the beginning of the research procedure until the baby is positioned will be excluded from the study. Instead of excluded infants, the first infant who met the inclusion criteria of the study and presented to the emergency department will be included.
* Bladder stimulation technique will not be applied.
* The infant will be evaluated by the observers at the 1st and 3rd minutes with the FLACC pain scale.
* Heart rate and saturation will be recorded at the 1st and 3rd minutes.
* The success of the procedure and the duration of the procedure will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Collecting urine specimen
* Between 1-12 months
* Being fed orally
* Having written consent from parents
* Complete skin integrity in the area where the maneuver will be performed

Exclusion Criteria:

* Poor general clinical condition (respiratory distress, etc.)
* Having signs of dehydration
* Having a diagnosed chronic health problem
* Having neurological and anatomical anomalies that may affect bladder function
* Any condition (intussusception, appendicitis, etc.) that will prevent the implementation of the stimulation maneuver.

Ages: 4 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedural success | During the procedure (3 minutes)
  Procedural success is defined as urine sample collection within 3 minutes (180 seconds) of starting the stimulation maneuvers.
Duration of the procedure | During the procedure (3 minutes)
  Duration of the procedure is defined as the time from the beginning of bladder stimulation to the beginning of micturition.

SECONDARY OUTCOMES:
Pain severity | Baseline (Before the procedure), at the 1st and 3rd minutes
  The pain levels of the infants during the procedure will determined by the researcher and a nurse who is a specialist in pediatric nursing by using the scale.
Heart rate | Baseline (Before the procedure), at the 1st and 3rd minutes
  The heart rate of the infants will measured with hand portable pulse oximeter
Peripheral oxygen saturation level | Baseline (Before the procedure), at the 1st and 3rd minutes
  The peripheral oxygen saturation levels of the infants will measured with hand portable pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Mutlu, Ph.d, Principal Investigator — Istanbul University - Cerrahpasa; Sinem Oral Cebeci, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Nihan Korkmaz, Şişli, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Altuntas N, Tayfur AC, Kocak M, Razi HC, Akkurt S. Midstream clean-catch urine collection in newborns: a randomized controlled study. Eur J Pediatr. 2015 May;174(5):577-82. doi: 10.1007/s00431-014-2434-z. Epub 2014 Oct 17. PMID 25319844
- [Background] Herreros Fernandez ML, Gonzalez Merino N, Tagarro Garcia A, Perez Seoane B, de la Serna Martinez M, Contreras Abad MT, Garcia-Pose A. A new technique for fast and safe collection of urine in newborns. Arch Dis Child. 2013 Jan;98(1):27-9. doi: 10.1136/archdischild-2012-301872. Epub 2012 Nov 21. PMID 23172785
- [Background] Kaufman J. How to... collect urine samples from young children. Arch Dis Child Educ Pract Ed. 2020 Jun;105(3):164-171. doi: 10.1136/archdischild-2019-317237. Epub 2019 Aug 23. PMID 31444213
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Morello W, La Scola C, Alberici I, Montini G. Acute pyelonephritis in children. Pediatr Nephrol. 2016 Aug;31(8):1253-65. doi: 10.1007/s00467-015-3168-5. Epub 2015 Aug 4. PMID 26238274
- [Background] Tran A, Fortier C, Giovannini-Chami L, Demonchy D, Caci H, Desmontils J, Montaudie-Dumas I, Bensaid R, Haas H, Berard E. Evaluation of the Bladder Stimulation Technique to Collect Midstream Urine in Infants in a Pediatric Emergency Department. PLoS One. 2016 Mar 31;11(3):e0152598. doi: 10.1371/journal.pone.0152598. eCollection 2016. PMID 27031953
- [Background] Şenaylı Y, Özkan F, Şenaylı A. Evaluation of postoperative pain in Turkish Translation. Turkish Clinics Journal of Anesthesiology Reanimation. 2006; 4(1): 1-4.